CLINICAL TRIAL: NCT04440657
Title: Self-assured Parents - a Parenting Support Program for Immigrant Parents With Teenage Children Living in Deprived Areas
Acronym: SAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University West, Sweden (Other)
Collaborators: Göteborg University (Other); Swedish Council for Working Life and Social Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020-01349
Record Dates: First submitted 2020-06-09; First posted 2020-06-19 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2023-12

CONDITIONS: Parenting; Parent-Child Relations; Adolescent Behavior
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immigrant parents (Experimental): All enrolled parents will be included in the parenting program
  Interventions: Behavioral: Self-Assured Parenting program

INTERVENTIONS:
Behavioral: Self-Assured Parenting program — Parents will receive parenting education for 10 weeks

SUMMARY:
Parents have the primary responsibility for child socialization and development, but not all parents have the same possibilities to promote their children's positive development. Immigrant parents living in deprived areas often worry about their children's safety and future, at the same time as they have difficulties facilitating the best development potential for their children. Social services can help parents and their children to attain more promising developmental outcomes through focus on early preventive parenting support efforts, but these efforts need to be culturally tailored for the best possible results. For this reason, social services in the municipality of Örebro developed a culturally sensitive parenting support program aimed at immigrant parents living in deprived areas, who are worried that their children (age 12-18) engage in or will be exposed to harmful environments.

The Self-Assured Parenting Program (SAP) offers support to these parents by building on protective factors and strengthening parents in their parenting through focus on parenting competence and parent-child communication.

The purpose of SAP is to increase parents' self-confidence and communication between parents and their teenagers as well as to reduce parents' worries through activities that have a clear focus on empowerment and knowledge of child development. This multi-design project aims to test the implementation and effect of TF in Örebro and other Swedish municipalities with similar problems through observation, interviews with parents and groupleaders/managers as well as longitudinal effect measurements of parenting competence, parent-child communication and worries about their children's psychosocial development. This project will allow a partnership between social workers and researchers to be formed in order to generate practice-based evidence about implementation of support to deprived parents, which can be used in the context of everyday social service practice.

ELIGIBILITY:
Inclusion Criteria:

* parents of adolescent Children
* immigrant background

Exclusion Criteria:

* parents of younger Children
* Swedish background

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Parent-child communication | 6 months
  Parent-child communication (Kerr & Stattin, 2000) will be assessed at 7 time points using an instrument with 22 questions measuring 1) Parent knowledge of child whereabouts (6 items) (e.g. "Do you know what places the child visits when he/she is out with his friends in the evenings?") 2) Parent control (5 items) (e.g. "Does the child need permission to stay out late on a weekday evening?") 3) Parent solicitation (6 questions) (e.g. "Do you ask the child to tell you about things that happen in his/her spare time?") and C hild Disclosure (5 items) (e.g. "When the child has been out one evening, does he/she want to tell you about what she/he has done?"). A 5-point Likert scale (1 - almost never to 5 - very often) will be used.
Change in Parents' worries | 6 months
  Parents' worries (Van Zalk et al., 2018) about their children will be assessed at 7 time points on a scale comprising six questions (e.g. "Are you worried that your child will get caught by the police?") answered on a 5-point Likert scale (1 - yes, always to 5 - no, never).
Change in Parental Self-efficacy | 6 months
  Parental self-efficacy will be assessed at 7 time points by the Parenting Sense of Competence in Parenting Scale (PSOC , Gilmore
  & C uskelly, 2009; Osman, 2017). The scale has subscales measuring satisfaction in parenting (9 items) (e.g.
  "Although parenting can be rewarding, I am frustrated now that the child is the age he/she is") and parental selfefficacy (7 items) (e.g. " I think I have what it takes to be a good parent to my child"). Answers are provided on 6-point Likert scales (1 - fully agree to 6 - completely disagree).

CONTACTS AND LOCATIONS:
Locations (1):
- University West, Trollhättan, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No